CLINICAL TRIAL: NCT01709617
Title: Sucrose as a Preferred Carbohydrate in Sports Nutrition
Brief Title: Carbohydrate Use During and Following Exercise
Acronym: CHO-use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 12-3-048
Record Dates: First submitted 2012-10-11; First posted 2012-10-18 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Carbohydrate Oxidation and Glycogen Utilization During and Following Exercise
Keywords: carbohydrate, glycogen, glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glucose-glucose (Experimental): Glucose ingestion
  Interventions: Dietary Supplement: Carbohydrate ingestion
- Glucose-Fructose (Active Comparator): glucose-fructose ingestion
  Interventions: Dietary Supplement: Carbohydrate ingestion
- disaccharide (Active Comparator): Disaccharide ingestion
  Interventions: Dietary Supplement: Carbohydrate ingestion

INTERVENTIONS:
Dietary Supplement: Carbohydrate ingestion — Various types of carbohydrate ingested during and following exercise

SUMMARY:
Carbohydrates are an integral component of sports nutrition. Providing carbohydrate (CHO) during exercise delays the onset of fatigue and improves exercise performance by maintaining high rates of CHO oxidation. Traditionally, glucose, or glucose polymers have been the preferential CHO source found in sports drinks. However, during the intestinal absorption of large amounts of glucose (>1.2 g/min), sodium-dependent glucose transporters (SGLT1) may become fully saturated, potentially limiting the rate of exogenous CHO oxidation. In an effort to evade this limitation, research has suggested using multiple transportable carbohydrates in the composition of sports drinks. Multiple transportable carbohydrates are combinations of simple sugars that use different intestinal transporters during the absorption process. Ingesting multiple transportable carbohydrates may enhance the capacity for total intestinal CHO absorption, leading to an increase in the rate of exogenous CHO oxidation. Our purpose will be to examine the disaccharide sucrose in it's ability to provide exogenous fuel during and following prolonged exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male
* 18 - 40 years of age
* Endurance trained cyclist/triathlete
* VO2 max ≥ 50 ml/kg/min
* BMI < 25 kg/m2

Exclusion Criteria:

* Use of medication
* Smoking

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-09 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Exogenous carbohydrate oxidation rate (Part A) | 0 min during trials 1-3
  Carbohydrate oxidation as measured by breath samples
Endogenous carbohydrate oxidation (Part A) | 0 min during trials 1-3
  endogenous carbohydrate oxidation as measured through breath samples during trials 1-3
Glycogen utilization (Part B) | immediately post exercise (~90min), during trials 4-6
  Glycogen utilization measured through a muscle biopsy sample at post (~90 min), 3 and 6 h post exercise.
  Part B; trials 4-6.
Exogenous carbohydrate oxidation rate (Part A) | 30 min during trials 1-3
  Carbohydrate oxidation as measured by breath samples
Exogenous carbohydrate oxidation rate (Part A) | 60 min during trials 1-3
  Carbohydrate oxidation as measured by breath samples
Exogenous carbohydrate oxidation rate (Part A) | 90 min during trials 1-3
  Carbohydrate oxidation as measured by breath samples
Exogenous carbohydrate oxidation rate (Part A) | 120 min during trials 1-3
  Carbohydrate oxidation as measured by breath samples
Exogenous carbohydrate oxidation rate (Part A) | 150 min during trials 1-3
  Carbohydrate oxidation as measured by breath samples
Exogenous carbohydrate oxidation rate (Part A) | 180 min during trials 1-3
  Carbohydrate oxidation as measured by breath samples
Endogenous carbohydrate oxidation (Part A) | 30 min during trials 1-3
  endogenous carbohydrate oxidation as measured through breath samples during trials 1-3
Endogenous carbohydrate oxidation (Part A) | 60 min during trials 1-3
  endogenous carbohydrate oxidation as measured through breath samples during trials 1-3
Endogenous carbohydrate oxidation (Part A) | 90 min during trials 1-3
  endogenous carbohydrate oxidation as measured through breath samples during trials 1-3
Endogenous carbohydrate oxidation (Part A) | 120 min during trials 1-3
  endogenous carbohydrate oxidation as measured through breath samples during trials 1-3
Endogenous carbohydrate oxidation (Part A) | 150 min during trials 1-3
  endogenous carbohydrate oxidation as measured through breath samples during trials 1-3
Endogenous carbohydrate oxidation (Part A) | 180 min during trials 1-3
  endogenous carbohydrate oxidation as measured through breath samples during trials 1-3
Glycogen utilization (Part B) | 3 h post exercise during trials 4-6
  Glycogen utilization measured through a muscle biopsy sample at post (~90 min), 3 and 6 h post exercise.
  Part B; trials 4-6.
Glycogen utilization (Part B) | 6 h post exercise during trials 4-6
  Glycogen utilization measured through a muscle biopsy sample at post (~90 min), 3 and 6 h post exercise.
  Part B; trials 4-6.

SECONDARY OUTCOMES:
Indirect calorimetry (Part A) | every 30 min up to 180 min during trials 1-3
  Measurements of VO2, VCO2 and RER through indirect calorimetry measured every 30 minutes during trials 1-3
Plasma glucose | every 30 min up to 180 min during trials 1-6
  Plasma glucose measurements
Plasma insulin | every 30 minutes up to 180 min during trials 1-6
  plasma insulin measurements

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, Ph.D., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands